CLINICAL TRIAL: NCT07061262
Title: The Comparison of Postoperative Analgesic Efficacy Between External Oblique Plane Block and Subcostal Tap Block in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: External Oblique Plane Block and Subcostal Tap Block for Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 266-2023
Record Dates: First submitted 2025-06-23; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Peripheral Nerve Block; Cholecystectomy, Laparoscopic; Pain After Surgery
Keywords: Laparoscopic cholecystectomy; postoperative pain; subcostal plane block; external oblique intercostal plane block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No peripheral nerve block
- External Oblique Plane Block (Experimental): Right after general anaesthesia induction and patient intubation, the patient will be placed in a supine position. Following sterile skin preparation, an external oblique plane block will be performed by the same anaesthesiologist under ultrasound guidance, using an external oblique muscle approach, in addition to standard analgesia applied in the control group.
  Interventions: Procedure: External Oblique Intercostal Plane Block
- Subcostal Plane Block (Active Comparator): Right after general anaesthesia induction and patient intubation, the patient will be placed in a supine position. Following sterile skin preparation, a subcostal block will be performed by the same anaesthesiologist under ultrasound guidance with subcostal approach, in addition to standard analgesia applied in the control group.
  Interventions: Procedure: Subcostal TAP block and spinal anesthesia group (STAP)

INTERVENTIONS:
Procedure: External Oblique Intercostal Plane Block — Right after general anaesthesia induction and patient intubation, the patient will be placed in a supine position. Following sterile skin preparation, an external oblique plane block will be performed by the same anesthesiologist under ultrasound guidance, using an external oblique muscle approach. A 22-gauge, 50-mm insulated stimulating needle will be used to administer 20 mL of anaesthetic solution (0.25% bupivacaine, 20 mL). Finally, 20 mL of local anaesthetic solution (0.25% bupivacaine anaesthetic solution) will be administered to disperse within the external oblique space.
  Arms: External Oblique Plane Block
Procedure: Subcostal TAP block and spinal anesthesia group (STAP) — Right after general anaesthesia induction and patient intubation, the patient will be placed in a supine position. Following sterile skin preparation, a subcostal block will be performed by the same anaesthesiologist under ultrasound guidance with a subcostal approach. A 22-gauge, 50-mm insulated stimulating needle will be used to administer 20 mL of anaesthetic solution (0.25% bupivacaine, 20 mL). Finally, 20 mL of local anaesthetic solution (0.25% bupivacaine anaesthetic solution) will be administered to disperse within the subcostal space.
  Arms: Subcostal Plane Block

SUMMARY:
The study aims to compare the efficacy of the external oblique plane block and the subcostal plane block in providing pain relief during perioperative anaesthetic management. As intraoperative haemodynamic stability is an important factor for surgeons to achieve better outcomes due to its effect on the quality of laparoscopic intervention, the investigator will observe its impact on this matter.

Ninety patients scheduled for elective surgery will be randomly assigned by a closed-envelope method into three groups (n = 30) receiving either a subcostal plan block, an external oblique plane block, or a control block preoperatively. Each group receive standardised general anaesthesia and perioperative pain management protocol. The data to be recorded include a numeric rating scale, intraoperative and postoperative analgesic use, intraoperative haemodynamic parameters, and VAS score. Moreover, block performance time, motor block and side effects or complications will be noted.

DETAILED DESCRIPTION:
All patients will receive standard general anaesthesia under standard monitorization; induction with 0,1-0,4 mg/kg midazolam, 2-2,5 mg/kg propofol, 1-2 mcq/kg fentanyl, 0,6-1,0 mg /kg rocuronium followed by 2% MAC sevoflurane in an air-oxygen mixture for maintenance of anaesthesia. Randomization is designed with concealed opaque envelope in a 1:1 ratio into two block groups (n= 30): subcostal plane block (Group A) and external oblique plane block (Group B) and control group ( Group C ). All blocks will be performed before surgical incision by a single experienced regional anaesthesiologist (A.A.) under ultrasound guidance with same local anaesthetic doses: 0.25% bupivacaine anaesthetic solution of 20 ml. The anaesthesia technician will record the duration of the block procedure. Then the investigator will apply dexamethasone 8 mg (IV), NSAIDs and after the patient will be ready for surgical incision. Intraoperative haemodynamic values (heart rate, systolic and mean arterial pressure) will be recorded by the same technician. The same analgesia protocol will be applied, consisting of an infusion of remifentanil (0.01 to 0.1 μg · kg-1 · min-1) if only needed to maintain heart rate and mean blood pressure within 20% of pre-induction values, and 1 g of paracetamol. Pain will be evaluated using both a numeric rating scale (0-10) and a verbal rating scale, starting at the post-anaesthesia care unit (PACU) and at time intervals of 2, 6, 12, and 24 hours postoperatively. Patients with persistent pain scores of higher than 4 out of 10 will receive rescue analgesia with 1mg/kg (maximum daily dose, 4x1) tramadol and 1 g (maximum daily dose, 4x1) paracetamol.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) Physical Status classification I to III

  * Patients who will give informed consent to peripheral nerve blocks

Exclusion Criteria:

* Refusal to participate in the study
* History of neurologic deficits or neuropathy
* Infection at the site of the block application
* Coagulopathy
* bleeding disorders
* Allergy to local anaesthetics
* Uncooperative patients who cannot reliably respond to verbal pain evaluation
* Kidney Failure
* Liver Failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Pain Score | postoperative day 1
  Numeric rating scale (NRS) worst pain imaginable as 10 points to zero for no pain.

SECONDARY OUTCOMES:
The total amount of analgesic drugs used | postoperative day 1
  The total amount of analgesic drugs used during the postoperative follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Berna Caliskan, Study Director — Haseki Training and Research Hospital: Istanbul Haseki Egitim Ve Arastirma Hastanesi
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kar S, Agrawal H, Yelamanchi R, Jain A, Kumar A, Agarwal N, Gupta N. Laparoscopy-guided transverse abdominis plane block versus port site infiltration for post-operative pain relief after laparoscopic cholecystectomy. J Minim Access Surg. 2025 Apr 1;21(2):126-132. doi: 10.4103/jmas.jmas_242_23. Epub 2024 Jul 30. PMID 39095984
- [Background] Qi-Hong S, Xu-Yan Z, Xu S, Yan-Jun C, Ke L, Rong W. Comparison of Ultrasound-Guided Erector Spinae Plane Block and Oblique Subcostal Transverse Abdominis Plane Block for Postoperative Analgesia in Elderly Patients After Laparoscopic Colorectal Surgery: A Prospective Randomized Study. Pain Ther. 2021 Dec;10(2):1709-1718. doi: 10.1007/s40122-021-00329-x. Epub 2021 Oct 15. PMID 34652717
- [Background] Gangadhar V, Gupta A, Saini S. Comparison of analgesic efficacy of combined external oblique intercostal and rectus sheath block with local infiltration analgesia at port site in patients undergoing laparoscopic cholecystectomy: a randomized controlled trial. Anesth Pain Med (Seoul). 2024 Jul;19(3):247-255. doi: 10.17085/apm.24002. Epub 2024 Jul 31. PMID 39118335